CLINICAL TRIAL: NCT01589666
Title: Safety Study of Spray-Dried Solvent/Detergent-Treated Plasma for Infusion in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Entegrion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSX-102
Record Dates: First submitted 2011-08-02; First posted 2012-05-02 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Coagulation Defects
Keywords: Entegrion; Spray-dried Solvent/Detergent Plasma; Fresh Frozen Plasma; Transfusion; Resuscitation; Hemorrhage; Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spray-dried S/D-treated plasma (Experimental): Resusix (Spray-Dried Solvent/Detergent-Treated Plasma) uses source plasma from U.S.-licensed facilities as the starting material. Source plasma donors are selected from the AB blood type, which is considered a "universal" product.
  Interventions: Biological: Spray-dried S/D-treated Plasma; Drug: Spray-dried S/D-treated plasma

INTERVENTIONS:
Biological: Spray-dried S/D-treated Plasma — Infusion of 100 mL Spray-dried S/D-treated Plasma
  Other Names: Resusix
Drug: Spray-dried S/D-treated plasma — Infusion of 200mL Spray-dried S/D-treated plasma
  Other Names: Resusix
Biological: Spray-dried S/D-treated Plasma — Infusion of 500 mL Spray-dried S/D-treated plasma
  Other Names: Resusix
Biological: Spray-dried S/D-treated Plasma — Infusion of 750 mL Spray-dried S/D-treated Plasma
  Other Names: Resusix
Biological: Spray-dried S/D-treated Plasma — Infusion of 800 mL Spray-dried S/D-treated Plasma
  Other Names: Resusix

SUMMARY:
This study is a Phase 1, single-center, open-label, ascending dose study which will assess the safety and tolerability of 5 doses of spray-dried solvent/detergent treated plasma (Resusix®) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent for participation in this study and valid contact information.
2. Subject must be a male or postmenopausal female.
3. Subject must be at least 18 years of age and not older than 55 years of age.
4. Subject must be in good general health, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening, including no history or symptoms of respiratory or cardiac disease.
5. Vital signs should be within normal limits at Screening:

   1. Body temperature within 97°F to 99°F
   2. Heart rate 45 to 100 beats per minute (bpm)
   3. Systolic blood pressure (SBP) within 90 to 140 mmHg and DBP within 50 to 90 mmHg.
6. Subject must have a normal (no clinically significant abnormality) EKG at Screening and prior to administration of Resusix

   1. PR interval within 120 and 200 mm/s
   2. QRS interval <120 mm/s
   3. QTc interval ≤440 mm/s
7. Subject must have laboratory hematology values within following normal ranges:

   1. White blood cell count (WBC): 4,500 to 11,000/mL
   2. Platelet (PLT) count: 150,000 to 400,000/mL;
   3. Hemoglobin (Hb): 12.5 to 15.5 g/dL;
   4. Activated partial thromboplastin time (aPTT): 24.6 to 36.7 seconds;
   5. Normal PT, International Normalized Ratio (INR): 0.8 to 1.2;
   6. Protein C ≥90%, Protein S ≥77%;
   7. Antithrombin III levels (ATIII) ≥100%.
8. Subject must have laboratory clinical chemistry values within normal range specified by the testing laboratory.
9. BMI ≤30 kg/m2.
10. Subject must have a negative toxicology screening panel (urine test including qualitative identification of PCP, barbiturates, THC, amphetamines, benzodiazepines, opiates, and cocaine.)
11. Subject must be a non-drinker (≤2 alcoholic beverages per week) and a non-smoker (any tobacco products within six months prior to Screening).
12. Subject must have no history of recreational (including IV) drug use (by self-declaration).
13. Subject must have the ability and willingness to attend frequent visits to the study center.

Exclusion Criteria:

1. Subject with lower extremity deep vein thrombosis (DVT) at Screening.
2. Subject has a history of coagulopathy or thromboembolic disease.
3. Subject has a first degree family member with history of venous thromboembolic disease <55 years of age or arterial thromboembolic disease <45 years of age.
4. Subject has documented drug allergies with well-described reactions.
5. Subject has hepatomegaly, splenomegaly, adenopathy, bruising, and/or ecchymoses identified at Screening.
6. Subject is found to have positive NAT test for HIV, HBV or HCV.
7. Subject has any murmurs, rubs, or gallops on cardiac auscultation.
8. Subject has had a previous transfusion at any time.
9. Subject is unlikely to comply with the study protocol or, in the opinion of the investigator, would not be a suitable candidate for participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent SAEs | 12 weeks
  Incidence of treatment-emergent SAEs reported for up to 12 weeks post Resusix infusion

SECONDARY OUTCOMES:
Change from baseline of select coagulation factors | 30 minutes post infusion
  To evaluate the recovery of select coagulation factors after infusion of 2 Resusix
Incidence of AEs | 12 weeks
  To evaluate the incidence of AEs for up to 12 weeks after infusion of Resusix

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Vince, DO, Principal Investigator — Vince & Associates Clinical Research, Inc.
Locations (1):
- Vince & Associates Clinical Research, Overland Park, Kansas, United States